CLINICAL TRIAL: NCT06338579
Title: Overview and Determinants of Self-medication Among Personnel Deployed on French Navy Surface Ships
Brief Title: Overview of Self-medication Among French Navy Personnel
Acronym: AutoMMaN
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PPRC04; 2023-A01763-42 (Other: IDRCB)
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Self Medication
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — A questionnaire is distributed and self-administered 4 weeks before the start of an embarked mission on a surface ship at the Toulon naval base, during an embarked mission of at least 4 weeks.
  The questionnaire consists of 2 parts:
  * A section on socio-demographic characteristics
  * A section on self-medication practices during this deployment

SUMMARY:
The goal of this cross-sectional descriptive observational study is to assess the extent of self-medication among the crews of surface ships at the Toulon naval base. This study could include healthy volunteers, or participants with well-controlled chronic pathologies enabling them to be fit for embarkation, who are currently being deployed for at least 4 weeks on a surface ship at the naval base.

Participants will tick and complete a questionnaire (between 15 and 30 minutes) after 4 consecutive weeks on the ship.

ELIGIBILITY:
Inclusion Criteria:

* French military personnel;
* age > 18;
* embarked on a French navy vessel from the naval base;
* for a minimum 4-week mission;
* covered by social security.

Exclusion Criteria:

* Refusal to participate,
* Legionnaire
* Military Health Services member

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers, or participants with well-controlled chronic pathologies enabling them to be fit for embarkation, military personnel currently deployed for at least 4 weeks on a naval base surface ship
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
percentage of patients who have self-medication | up to 4 weeks
  Percentage of patients who have self-medicated at least once since the start of their current mission, among respondents working on surface ships at the naval base on missions lasting more than 4 weeks (excluding malaria prophylaxis, contraception and treatment of a chronic pathology prescribed by a doctor)

IPD SHARING:
Plan to Share IPD: No